CLINICAL TRIAL: NCT02936492
Title: Escalating Dose Study for Safety, Tolerability and Pharmacokinetics After Single and Multiple Dermal Administration of Two BAY1003803 Formulation Types With Two Concentrations Each in Healthy Male Volunteers, Applying a Double-blind, Vehicle-controlled Design and Including a Positive Control Group
Brief Title: BAY1003803 Single and Multiple Dose Escalation, Safety, Tolerability and Pharmacokinetics Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 17014
Record Dates: First submitted 2016-10-17; First posted 2016-10-18 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Psoriasis
Keywords: Phase I; Healthy volunteers
MeSH Terms: conditions — Psoriasis | interventions — Ointments; Clobetasol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAY1003803 (Experimental): Topical treatment: dose escalating in 9 steps from 0.13 mg to 61.7 mg per subject
  Interventions: Drug: BAY1003803 0.01% lipophilic cream; Drug: BAY1003803 0.1% lipophilic cream; Drug: BAY1003803 0.01% ointment; Drug: BAY1003803 0.1% ointment
- Placebo (Placebo Comparator): Topical treatment using matching amount of placebo
  Interventions: Drug: Lipophilic cream vehicle; Drug: Ointment vehicle
- Clobetasol propionate (Active Comparator): Topical treatment using 16.5 mg of clobetasol propionate per subject
  Interventions: Drug: Clobetasol propionate

INTERVENTIONS:
Drug: BAY1003803 0.01% lipophilic cream — Topical administration for 22 h per day
  Arms: BAY1003803
Drug: BAY1003803 0.1% lipophilic cream — Topical administration for 22 h per day
  Arms: BAY1003803
Drug: BAY1003803 0.01% ointment — Topical administration for 22 h per day
  Arms: BAY1003803
Drug: BAY1003803 0.1% ointment — Topical administration for 22 h per day
  Arms: BAY1003803
Drug: Lipophilic cream vehicle — Topical administration for 22 h per day
  Arms: Placebo
Drug: Ointment vehicle — Topical administration for 22 h per day
  Arms: Placebo
Drug: Clobetasol propionate — Topical administration for 22 h per day
  Arms: Clobetasol propionate

SUMMARY:
Systemic safety following single and multiple dermal administration of BAY1003803

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subject
* Age: 18 to 64 years (inclusive) at the first screening visit
* Body mass index (BMI): above or equal 18 and below or equal 30 kg / m² at the first screening visit
* Non-smoker at least 3 months prior to study start and during the study
* Healthy skin on which reddening can be easily recognized

Exclusion Criteria:

* A history of relevant diseases, especially incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, excretion and effect of the study drugs will not be normal, dermal diseases, diseases which present a risk for subjects to be treated with glucocorticoid receptor agonists (e.g. gastric ulcers, cornea ulcer, colitis ulcerosa, severe infections, glaucoma, diabetes, myocardial infarction, thromboembolic disease, hypertension, thyroid disease, tuberculosis, myasthenia gravis, osteoporosis, psychiatric diseases)
* Infections and febrile illness within 4 week before the first study drug administration
* Use of systemic or topical medicines or substances which oppose the study objectives or which might influence them
* Inoculations with live vaccine within 8 weeks before the first study drug administration
* Signs of irritation or folliculitis or any other dermatological conditions in the test areas that would interfere with the planned assessments as judged by the Investigators
* Human leukocyte antigen-DR (HLA-DR) < 15000 AB/monocyte

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-10-24 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Cortisol serum levels for safety | Up to 2 weeks
Frequency of treatment-emergent adverse events (TEAEs) | Up to 2 weeks
Nature of treatment-emergent adverse events (TEAEs) | Up to 2 weeks

SECONDARY OUTCOMES:
Monocytic human leukocyte antigen-DR (HLA-DR) expression (Part 1, single dose) | Day 1 to 3 at 8:00 am
Monocytic human leukocyte antigen-DR (HLA-DR) expression (Part 2, multiple dose) | Day 1 to 8 at 8:00 am
Maximum plasma concentration (Cmax) after single dose of BAY1003803 | At pre-dose, 1.5, 3, 5, 7, 9, 11, 13, 15, 21, 22, 23, 24 hours
Area under the plasma concentration vs. time curve from zero to infinity (AUC) after single dose of BAY1003803 | At pre-dose, 1.5, 3, 5, 7, 9, 11, 13, 15, 21, 22, 23, 24, 27, 31, 35, 39, 47 hours
Area under the curve from time zero to 22 hours [AUC(0-22)] after single dose of BAY1003803 | At pre-dose, 1.5, 3, 5, 7, 9, 11, 13, 15, 21, 22 hours
Maximum plasma concentration (Cmax,md) after multiple dose of BAY1003803 | At pre-dose, 3, 7, 9, 11, 13, 22, 23 hours (Day 1); At pre-dose, 3, 7, 9, 11, 13, 22, 23, 24 hours (Day 2 and Day 6)
Area under the curve from time zero to 24 hours [AUC(0-24)md] after multiple dose of BAY1003803 | At pre-dose, 3, 7, 9, 11, 13, 22, 23 hours (Day 1); At pre-dose, 3, 7, 9, 11, 13, 22, 23, 24 hours (Day 2 and Day 6)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Hamburg, Germany